CLINICAL TRIAL: NCT01302327
Title: GLP Analogs for Diabetes in Wolfram Syndrome Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Very rare disease, we were unable to recruit patients
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Adar Zinger, Physician, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: wolfram-HMO-CTIL
Record Dates: First submitted 2011-02-22; First posted 2011-02-24 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Diabetes Mellitus Associated With Genetic Syndrome; Wolfram Syndrome
Keywords: Wolfram syndrome; Diabetes mellitus; Exenatide; GLP-1 analog; beta cell function
MeSH Terms: conditions — Wolfram Syndrome; Diabetes Mellitus | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exenatide (Experimental)
  Interventions: Drug: Exenatide

INTERVENTIONS:
Drug: Exenatide — Exenatide

SUMMARY:
Wolfram syndrome, also referred to as DIDMOAD (diabetes insipidus, diabetes mellitus, optic atrophy and deafness) is a genetic syndrome characterized by beta-cell dysfunction and apoptosis leading to diabetes, neurodegeneration and psychiatric illness. Accumulating evidence indicates that beta-cell failure and neuronal cell dysfunction in Wolfram's syndrome results from a high level of ER stress in affected cells. The current treatment of Wolfram syndrome is insulin, which fails to prevent the progression of beta-cell failure.

Several studies showed that GLP-1 analogs are very effective in protecting beta-cells from ER stress. Herein, the investigators suggest studying the impact of GLP-1 analogs in the treatment of patients with Wolfram syndrome.

The investigators will Study the effects of GLP-1 analog (Exanatide) on beta-cell function and glycemic control of patients with Wolfram syndrome. Evaluation of beta cell function will be done by performing meal test and IVGTT test before starting GLP-1 therapy, and after 3 month of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic or definitive clinical diagnosis of Wolfram's syndrome including: diabetes mellitus, optic atrophy and at least one additional neurological dysfunction (diabetes insipidus, sensorineural deafness, neurogenic bladder or other type of autonomic or peripheral neuropathy)
2. Age >18 years
3. Duration of diabetes of <10 years.

Exclusion Criteria:

1. pregnant women
2. patients who are unable to give inform consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03-01; Primary Completion 2013-03-01 (Estimated); Study Completion 2013-03-01 (Actual)

PRIMARY OUTCOMES:
beta cell function | 3 months
  IVGTT test and meal test will be performed before starting treatment with Exenetide and after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Gil Leibowitz, MD, Principal Investigator — Hadassah Medical Organization

REFERENCES:
- [Derived] Danielpur L, Sohn YS, Karmi O, Fogel C, Zinger A, Abu-Libdeh A, Israeli T, Riahi Y, Pappo O, Birk R, Zangen DH, Mittler R, Cabantchik ZI, Cerasi E, Nechushtai R, Leibowitz G. GLP-1-RA Corrects Mitochondrial Labile Iron Accumulation and Improves beta-Cell Function in Type 2 Wolfram Syndrome. J Clin Endocrinol Metab. 2016 Oct;101(10):3592-3599. doi: 10.1210/jc.2016-2240. Epub 2016 Jul 26. PMID 27459537